CLINICAL TRIAL: NCT02048527
Title: Comparison of Single-step (Global) Versus Sequential Media (Origio) in Preimplantation Embryo Development and Pregnancy Rates
Brief Title: Single-step Versus Sequential Media in Preimplantation Embryo Development and Pregnancy Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Global versus Origio
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Global (Active Comparator): In vitro embryo culture in single-step medium (Global)
  Interventions: Other: Global
- Origio (Active Comparator): In vitro embryo culture in sequential media (Origio)
  Interventions: Other: Origio

INTERVENTIONS:
Other: Global — Single medium for the culture of embryos from Day1 to Day 5
  Other Names: Global medium (LIfeGlobal)
  Arms: Global
Other: Origio — Sequential media medium for the culture of embryos from Day1 to Day 3 (ISM1) and from Day 3 to Day 5 (BlastAssist)
  Other Names: ISM1/BlastAssist (Origio)
  Arms: Origio

SUMMARY:
Sequential culture media were introduced in order to meet the changing requirements of the developing embryo in vitro. However, there has been renewed interest in the use of single-step media, which allow the embryo itself to choose the necessary nutrients while maintaining a more stable culture environment. Previous studies suggest that sequential media do not appear superior to single-step media.

DETAILED DESCRIPTION:
Sequential culture media were introduced in order to meet the changing requirements of the developing embryo in vitro. However, there has been renewed interest in the use of single-step media, which allow the embryo itself to choose the necessary nutrients while maintaining a more stable culture environment. Previous studies suggest that sequential media do not appear superior to single-step media.

The current study will include 2 RCTs:

RCT 1: Random allocation of sibling oocytes to compare embryo development and blastocyst formation rates in the two culture media compared.

RCT2: Random allocation of patients in either Global or Origio media, to evaluate pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* <40 years of age
* female infertility patients
* at least 10 retrieved oocytes

Exclusion Criteria:

* 41 years or older
* frozen-thawed oocytes/embryos
* oocyte donation cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Implantation rate per embryo transferred | 7 weeks
  Number of fetal sacs with positive heart beat at 7 weeks of gestation

SECONDARY OUTCOMES:
Blastocyst formation rate | Day 5
  Embryos reaching the blastocyst stage on Day 5 post oocyte retrieval
Good quality blastocysts | Day 5
  Good quality blastocysts are considered at least full blastocysts (stage 3 and above) with grade A or grade B inner-cell mass and trophectoderm respectively.
Positive hCG rates | 14 days
  Pregnancy test as assessed by detection of hCG using blood test
Ongoing pregnancy rates | 12 weeks
  Pregnancy reaching 12 weeks of gestation
Early pregnancy loss | 12 weeks
  Miscarriage per positive hCG test up to 12 weeks of gestation
Clinical pregnancy | 7 weeks
  Pregnancy reaching 7 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis A Sfontouris, PhD, Principal Investigator — Eugonia; Trifon G Lainas, PhD, Study Director — Eugonia
Locations (1):
- Eugonia Assisted Reproduction Unit, Athens, Attica, Greece

REFERENCES:
- [Background] Sepulveda S, Garcia J, Arriaga E, Diaz J, Noriega-Portella L, Noriega-Hoces L. In vitro development and pregnancy outcomes for human embryos cultured in either a single medium or in a sequential media system. Fertil Steril. 2009 May;91(5):1765-70. doi: 10.1016/j.fertnstert.2008.02.169. Epub 2008 Apr 25. PMID 18439587
- [Background] Basile N, Morbeck D, Garcia-Velasco J, Bronet F, Meseguer M. Type of culture media does not affect embryo kinetics: a time-lapse analysis of sibling oocytes. Hum Reprod. 2013 Mar;28(3):634-41. doi: 10.1093/humrep/des462. Epub 2013 Jan 12. PMID 23315059